CLINICAL TRIAL: NCT01388829
Title: A Phase 1, Single-Dose, Open-Label, Crossover Study To Assess The Relative Bioavailability Of 2 Different Formulations Of PF-04991532
Brief Title: Study To Assess The Pharmacokinetics Of 2 Different Formulations Of PF-04991532
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B2611015
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: formulation comparison

ARMS (1):
- formulation comparison (Experimental): formulation comparison
  Interventions: Drug: Treatment A; Drug: Treatment B

INTERVENTIONS:
Drug: Treatment A — 150 mg single dose of PF 04991532 tablets (1x150 mg) manufactured from the R3 lot
Drug: Treatment B — 150 mg single dose of PF 04991532 tablets (1x150 mg) manufactured from the R4 lot

SUMMARY:
This study is designed to compare the pharmacokinetics of two different lots of tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non childbearing potential) subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests. Women must be of non childbearing potential as defined in Lifestyle Guidelines.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject or a legally acceptable representative.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at Screening.
* Screening supine blood pressure 140 mm Hg (systolic) or 90 mm Hg (diastolic), on a single measurement [confirmed by a single repeat, if necessary] following at least 5 minutes of rest.
* Any condition possibly affecting drug absorption (eg, gastrectomy).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Plasma AUClast | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours
Plasma Cmax | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours

SECONDARY OUTCOMES:
Plasma Tmax | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2611015&StudyName=Study%20To%20Assess%20The%20Pharmacokinetics%20Of%202%20Different%20Formulations%20Of%20PF-04991532